CLINICAL TRIAL: NCT01581554
Title: Withdrawal of Therapy After Long-Term Oral Nucleos(t)Ide Analogue Treatment in Patients With Chronic Hepatitis B
Brief Title: Withdrawal of Therapy After Long-Term Antiviral Treatment for Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110151; 11-DK-0151
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-04-15

CONDITIONS: Chronic Hepatitis B e Antigen Positive; Chronic Hepatitis B e Antigen Negative
Keywords: Hepatitis B; Treatment; Nucleoside/Nucleotide Analogue; Natural History
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with HBeAg negative chronic hepatitis B: Patients with HBeAg negative chronic hepatitis B who have received a minimum of 4 years of oral nucleoside therapy with a serum HBV DNA level less than 500 IU/ml in the 6 months prior to withdrawal.
- Patients with HBeAG positive chronic hepatitis B: Patients with HBeAg positive chronic hepatitis B who have received a minimum of 4 years of oral nucleoside therapy with a serum HBV DNA level less than 500 IU/ml in the 6 months prior to withdrawal.

SUMMARY:
Background:

- Chronic infection with the hepatitis B virus may lead to cirrhosis, liver disease, and cancer of the liver. There is no cure for the infection, but several drugs have been approved to treat it. These drugs can keep the virus levels low. They seem to be safe for short-term use. But the drugs have not yet been approved for long-term use because some of them can have serious side effects. However, stopping treatment too soon can make the infection worse and may lead to more serious forms of liver disease. Researchers have not been able to determine a when to stop treatment. They want to study people with chronic hepatitis B infection to find out the best time to stop treatment and prevent the disease from causing further liver damage.

Objectives:

* To study the safety and effectiveness of withdrawing antiviral treatment for chronic hepatitis B after at least 4 years of treatment.
* To determine whether stopping long-term antiviral treatment for chronic hepatitis B makes the infection worse.

Eligibility:

- People who are at least 18 years of age; have been taking antiviral drugs to treat chronic hepatitis B for at least 4 years; and are being evaluated to stop treatment.

Design:

* Those in the study will be screened with a physical exam, medical history, questionnaire, and blood tests. They will remain under the care of their regular doctor during the study.
* They will have an abdominal ultrasound to study scarring in the liver, if they have not had one in the past year.
* Those without detectable levels of the hepatitis B virus in their blood will stop antiviral treatment. They will have monthly blood tests for the first 6 months to check virus levels, and then every 3 months afterward.
* Those whose blood tests show an increase in virus levels will restart antiviral treatment as directed by the study doctors and their personal doctor.
* All those in the study will be monitored until the end of the study.

DETAILED DESCRIPTION:
Chronic hepatitis B affects at least 1.5 million Americans and is a major cause of cirrhosis, end-stage liver disease and hepatocellular carcinoma. Five oral antiviral agents have been licensed for use in chronic hepatitis B in the United States. These agents are effective at suppressing viral replication, improving liver disease and reversing cirrhosis. The standard indications for starting antiviral therapy have been developed and widely accepted. Less clear is how long therapy should continue and when and under what conditions should therapy be stopped. Withdrawal after one year of therapy is commonly followed by relapse that in rare instances is severe and can be fatal. With longer courses of therapy, withdrawal of antiviral therapy has been associated with fewer and less severe relapses, but the criteria for stopping treatment are still unclear.

In this study, we propose to withdraw therapy in up to 50 patients with both HBeAg positive and negative chronic hepatitis B who have received a minimum of 4 years of oral nucleoside therapy with a serum HBV DNA level less than 500 IU/ml in the 6 months prior to withdrawal. After an outpatient evaluation, consenting patients will be withdrawn from therapy and followed carefully for presence of symptoms, abnormal liver tests and HBV DNA levels monthly for 6 months and every 3 months thereafter. Patients who relapse will be offered retreatment. Patients without relapse will be followed for at least four years after stopping therapy. The primary endpoint of the study will be the proportion of patients who maintain an HBV DNA < 1,000 IU/ml, and a serum ALT or AST<1.5 times the upper limit of normal one year off therapy. Secondary endpoints will be the proportion of patients who maintain HBeAg loss and clear HBsAg one year off therapy, the number of ALT or AST flares, predictors of maintained virological suppression and HBeAg negativity and the proportion of subjects who require re-initiation of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 18 years and older, male or female

HBsAg positive for greater than 6 months

For HBeAg positive subjects, HBeAg loss with or without anti-HBe with a minimum period of antiviral therapy for 48 weeks after HBeAg loss was first detected.

HBV DNA less than or equal to 500 IU/mL tested on at least 2 occasions over the last 6 months

Antiviral therapy for a minimum of 4 years

Baseline ALT or AST within the upper limit of normal.

Willing and able to provide written, informed consent.

Subjects must be eligible to enter protocol 07-DK-0207 or be willing to be treated by their local physician should relapse or a hepatitis flare occur.

EXCLUSION CRITERIA:

Presence of cirrhosis (Ishak fibrosis score 5 or 6) on any liver biopsy performed within the last 4 years. In the absence of a liver biopsy then any three of the following five variables: platelet count less than or equal to 100,000/mm(3), reversal of ALT/AST ratio, total bilirubin greater than 2.0 mg/dL, splenomegaly on ultrasound and presence of esophageal or gastric varices or portal hypertensive gastropathy on endoscopy

Any history of decompensated liver disease

Prior or current therapy with tenofovir or tenofovir plus emtricitabine

Renal insufficiency defined as a serum creatinine greater than 1.5 mg/dL or an estimated glomerular filtration rate less than or equal to 50 mls/minute using the Cockroft and Gault formula.

Anti-hepatitis C virus positivity

Anti-hepatitis D virus positivity

Anti-human immunodeficiency virus positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver clinic population and community
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-05-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who maintain an HBV DNA <1.5 X the upper limit of normal one year off therapy | One year after stopping therapy
  Proportion of patients who maintain an HBV DNA <1,000 IU/ml, and a serum ALT or AST <1.5 X the upper limit of normal one year off therapy

SECONDARY OUTCOMES:
Proportion of patients who maintain HBeAg loss and clear HBsAg one year off therapy | One year after stopping therapy
  Proportion of patients who maintain HBeAg loss and clear HBsAg
Number of ALT or AST flares | One year after stopping therapy
  Number of ALT or AST flares

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-DK-0151.html